CLINICAL TRIAL: NCT05613205
Title: A Phase 1, Observer-blind, Randomised, Controlled, Single-centre Study to Evaluate the Safety, Reactogenicity, and Immune Responses to an Adjuvanted and Non-adjuvanted Conjugate Vaccine Against Salmonella Typhi and Salmonella Paratyphi A in Healthy Adults 18 to 50 Years of Age in Europe
Brief Title: Safety and Immunogenicity of a Novel Conjugate Vaccine Against Salmonella Typhi and Salmonella Paratyphi A in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Biological E. Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 205480; 2021-002029-19 (EudraCT Number)
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Typhoid Fever
Keywords: Salmonella Typhi; Salmonella Paratyphi A; Typhoid fever; Paratyphoid fever; Enteric fever; Conjugate vaccine; First-time-in-human
MeSH Terms: conditions — Typhoid Fever; Paratyphoid Fever | interventions — Adjuvants, Vaccine; Vaccines; Vi polysaccharide vaccine, typhoid; Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind (Day 1 to Day 29) and in a Single-blind (Day 29 to Day 337) manner with participants and investigator blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Step 1a: Low dose TYP04A vaccine without Alum (Experimental): Participants received low dose of the TYP04A vaccine without Alum intramuscularly on Day 1 and Day 169.
  Interventions: Biological: TYP04A Low Dose without Alum investigational vaccine
- Step 1b: Low dose TYP03A vaccine with Alum (Experimental): Participants received low dose of the TYP03A vaccine with Alum intramuscularly on Day 1 and Day 169.
  Interventions: Biological: TYP03A Low Dose with Alum investigational vaccine
- Step 2: Full dose TYP04B vaccine without Alum (Experimental): Participants received full dose of the TYP04B vaccine without Alum intramuscularly on Day 1 and day 169.
  Interventions: Biological: TYP04B Full Dose without Alum investigational vaccine
- Step 2: Full dose TYP03B vaccine with Alum (Experimental): Participants received full dose of the TYP03B vaccine with Alum intramuscularly on Day 1 and day 169.
  Interventions: Biological: TYP03B Full Dose with Alum investigational vaccine
- Control: TYPHIM VI and BOOSTRIX vaccine (Active Comparator): Participants received TYPHIM VI as comparator intramuscularly on Day 1, and BOOSTRIX as comparator on Day 169.
  Interventions: Biological: Sanofi Pasteur's Typhoid Vi polysaccharide vaccine; Biological: GSK's Tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine

INTERVENTIONS:
Biological: TYP04A Low Dose without Alum investigational vaccine — 2 doses of TYP04A Low Dose without Alum investigational vaccine administered intramuscularly as a priming dose on Day 1 and a booster dose on Day 169.
  Other Names: Typhoid and Paratyphoid A conjugate low dose without adjuvant vaccine
  Arms: Step 1a: Low dose TYP04A vaccine without Alum
Biological: TYP04B Full Dose without Alum investigational vaccine — 2 doses of TYP04B Full Dose without Alum investigational vaccine administered intramuscularly as a priming dose on Day 1 and a booster dose on Day 169.
  Other Names: Typhoid and Paratyphoid A conjugate full dose without adjuvant vaccine
  Arms: Step 2: Full dose TYP04B vaccine without Alum
Biological: TYP03A Low Dose with Alum investigational vaccine — 2 doses of TYP03A Low Dose with Alum investigational vaccine administered intramuscularly as a priming dose on Day 1 and a booster dose on Day 169.
  Other Names: Adjuvanted Typhoid and Paratyphoid A conjugate low dose vaccine
  Arms: Step 1b: Low dose TYP03A vaccine with Alum
Biological: TYP03B Full Dose with Alum investigational vaccine — 2 doses of TYP03B Full Dose with Alum investigational vaccine administered intramuscularly as a priming dose on Day 1 and a booster dose on Day 169.
  Other Names: Adjuvanted Typhoid and Paratyphoid A conjugate full dose vaccine
  Arms: Step 2: Full dose TYP03B vaccine with Alum
Biological: Sanofi Pasteur's Typhoid Vi polysaccharide vaccine — 1 dose of Sanofi Pasteur's Typhoid Vi polysaccharide vaccine administered intramuscularly, at Day 1, to participants in the control group.
  Other Names: TYPHIM VI
  Arms: Control: TYPHIM VI and BOOSTRIX vaccine
Biological: GSK's Tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine — 1 dose of GSK's Tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine administered intramuscularly, at Day 169, to participants in the control group.
  Other Names: BOOSTRIX
  Arms: Control: TYPHIM VI and BOOSTRIX vaccine

SUMMARY:
A bivalent Typhoid and Paratyphoid A conjugate investigational vaccine aimed to prevent both typhoid and paratyphoid enteric fever in infants and older age groups has been developed by GlaxoSmithKline (GSK).

The purpose of this first-time-in-human study is to evaluate the safety and immunogenicity profile of a low and a full dose of the investigational vaccine, formulated with or without adjuvant, administered in 2 doses, 24 weeks apart, in healthy adults 18 to 50 years of age in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the Investigator, can and will comply with the requirements of the Protocol (e.g., completion of the diary cards, return for follow-up visits).
* Written informed consent obtained from the participant prior to performance of any study specific procedure.
* Healthy participants as established by medical history, clinical examination, and screening laboratory investigations.
* Participant satisfying screening requirements.
* Participant seronegative for human immunodeficiency virus, hepatitis B, and hepatitis C at Screening.
* A male or female participant between, and including, 18 and 50 years of age at the time of the first study intervention administration.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the study intervention administration series.

Exclusion Criteria:

Medical conditions

* Progressive, unstable or uncontrolled clinical conditions.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Hypersensitivity, including allergy, to medicinal products or medical equipment whose use is foreseen in this study.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Any behavioural or cognitive impairment or psychiatric disease that, in the opinion of the Investigator, may interfere with the participant's ability to participate in the study.
* Acute* or chronic illness, clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by physical examination or laboratory screening tests.

  *Participants with a minor illness (such as mild diarrhoea or mild upper respiratory infection) without fever may be enrolled at the discretion of the Investigator.
* Any clinically significant* haematological and/or biochemical laboratory abnormality.

  *The Investigator should use his/her clinical judgement to decide which abnormalities are clinically significant.
* Confirmed positive COVID-19 test during the period starting 14 days before the first administration of study vaccines (Day -14 to Day 1).
* Any other clinical condition that, in the opinion of the Investigator, might pose additional risk to the participant due to participation in the study.
* Confirmed or suspected autoimmune diseases (e.g., vitiligo, autoimmune thyroiditis).

Prior/Concomitant therapy

* Previous administration of any type of Typhoid vaccine (Ty21a, Vi-PS, or Typhoid conjugate vaccine).
* Use of any investigational or non-registered product (drug, vaccine, or medical device) other than the study interventions during the period starting 30 days before the first administration of study vaccines (Day -30 to Day 1), or planned use during the study period.
* A vaccine not foreseen by the study protocol administered during the period starting at -14 days before the first dose (-21 days in the case of live vaccines) and ending 28 days after the last dose of study intervention administration*, with the exception of flu and COVID-19 vaccines, administered during the period starting at 7 days before and 7 days after each dose (14 days before and 14 days after in case of live vaccines).

  *In case emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is recommended and/or organised by public health authorities outside the routine immunisation programme, the time period described above can be reduced if, necessary for that vaccine, provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly. When regulations allow, the recommended time intervals for administration of these vaccines are at least 7 days before or 7 days after (at least 14 days before or 14 days after in case of live vaccines) each dose of study intervention administration.
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g., infliximab).
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the administration of the first dose of study intervention or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first study intervention dose. For corticosteroids, this will mean prednisone equivalent ≥20 mg/day for adult participants. Inhaled and topical steroids are allowed.

Prior/Concurrent clinical study experience • Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (drug/invasive medical device).

Other exclusions

* History of travel to countries of Asia that are considered endemic* for enteric fever in the last 3 years.

  *this also includes travel during study duration.
* Pregnant or lactating female.
* Female participants planning to become pregnant or planning to discontinue contraceptive precautions.
* History of or current chronic alcohol consumption and/or drug abuse.
* Any study personnel or immediate dependents, family, or household member.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] De Coster I, AbdelGhany M, Sarakinou E, Fineschi C, Marchetti E, La Gaetana R, Nigro S, Carducci M, Massai L, Conti V, Rossi O, Luna Cilio G, Serry-Bangura A, Tessitore P, Van Damme P, Withanage K, Micoli F, Berlanda Scorza F, Rondini S, Nakakana UN, Kumar Arora A. Safety and immunogenicity of a conjugate vaccine candidate against Salmonella enterica serovars Typhi and Paratyphi A in healthy adults in Europe: a phase 1 randomised controlled trial. Lancet Infect Dis. 2026 Jan 23:S1473-3099(25)00730-3. doi: 10.1016/S1473-3099(25)00730-3. Online ahead of print. PMID 41587557

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 97 participants enrolled, 1 participant, who underwent post-screening procedures, withdrew from the study before randomisation and did not receive the study intervention. Therefore, 96 participants were randomised in the study.
Groups:
- Step 1a: Low Dose TYP04A Vaccine Without Alum: Participants received a low dose of the TYP04A vaccine without Alum intramuscularly on Day 1 and Day 169.
- Control: TYPHIM VI and BOOSTRIX Vaccine: Participants received TYPHIM VI as the comparator intramuscularly on Day 1 and BOOSTRIX as the comparator on Day 169.
Period: Overall Study
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Started | 12 | 12 | 24 | 24 | 24
Completed | 12 | 12 | 22 | 22 | 24
Not Completed | 0 | 0 | 2 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population comprised of exposed set which included all participants who were assigned to study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine | Total
Number analyzed (Participants) | 12 | 12 | 24 | 24 | 24 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.9 (10.8) | 31.8 (8.4) | 27.0 (9.2) | 27.1 (9.8) | 30.7 (10.6) | 29.2 (9.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1 | 6 | 10 | 7 | 6 | 30
  Female | 11 | 6 | 14 | 17 | 18 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 12 | 24 | 24 | 24 | 96

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Administration-site Events After the First Vaccination
Description: Solicited administration site events included pain, redness, and swelling.
Time Frame: From Day 1 to Day 7
Population: The analysis was performed on the solicited safety set, which included all participants who received at least 1 dose of the study intervention and had solicited safety data during the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 12 | 23 | 24 | 24
Participants
  Pain | 3 | 11 | 20 | 22 | 17
  Redness | 1 | 0 | 1 | 1 | 0
  Swelling | 1 | 0 | 1 | 1 | 1

2. Primary Outcome: Number of Participants With Solicited Administration-site Events After the Second Vaccination
Description: Solicited administration site events included pain, redness, and swelling.
Time Frame: From Day 169 to Day 175
Population: The analysis was performed on the Solicited safety set. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 8 | 10 | 21 | 22 | 21
Participants
  Pain | 6 | 6 | 20 | 19 | 13
  Redness | 1 | 0 | 0 | 0 | 1
  Swelling | 1 | 0 | 2 | 1 | 0

3. Primary Outcome: Number of Participants With Solicited Systemic Events After the First Vaccination
Description: The solicited systemic events included arthralgia (joint pain), fatigue (tiredness), fever, headache, and myalgia (muscle pain). Fever is defined as body temperature more than or equal to (>=) 38.0 degrees Celsius (°C).
Time Frame: From Day 1 to Day 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 12 | 23 | 24 | 24
Participants
  Arthralgia | 1 | 3 | 2 | 2 | 2
  Fatigue | 4 | 3 | 9 | 12 | 11
  Fever | 0 | 0 | 0 | 1 | 0
  Headache | 5 | 5 | 10 | 6 | 11
  Myalgia | 3 | 3 | 7 | 15 | 9

4. Primary Outcome: Number of Participants With Solicited Systemic Events After the Second Vaccination
Description: The solicited systemic events included arthralgia (joint pain), fatigue (tiredness), fever, headache, and myalgia (muscle pain).
Time Frame: From Day 169 to Day 175
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 8 | 10 | 21 | 22 | 21
Participants
  Arthralgia | 0 | 1 | 1 | 2 | 3
  Fatigue | 1 | 3 | 6 | 9 | 9
  Fever | 0 | 0 | 0 | 0 | 0
  Headache | 2 | 3 | 9 | 9 | 9
  Myalgia | 3 | 3 | 9 | 9 | 9

5. Primary Outcome: Number of Participants With Unsolicited Adverse Events (AEs) After the First Vaccination
Description: An unsolicited AE is defined as an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Time Frame: From Day 1 to Day 28
Population: The analysis was performed on the unsolicited safety set, which included all participants who received at least 1 dose of the study intervention and reported having/not having unsolicited AEs during the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 12 | 24 | 24 | 24
Participants | 7 | 9 | 15 | 12 | 14

6. Primary Outcome: Number of Participants With Unsolicited Adverse Events After the Second Vaccination
Description: An unsolicited adverse event is defined as an adverse event that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events.
Time Frame: From Day 169 to Day 196
Population: The analysis was performed on the unsolicited safety set. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 8 | 10 | 21 | 22 | 21
Participants | 1 | 2 | 11 | 8 | 4

7. Primary Outcome: Number of Participants With Any Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, results in abnormal pregnancy outcomes or any other situation based on appropriate medical or scientific judgement.
Time Frame: From Day 1 to Day 197
Population: The analysis was performed on the exposed set, which included all participants who received at least 1 dose of the study intervention. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 12 | 24 | 24 | 24
Participants | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With AEs/SAEs Leading to Withdrawal From the Study
Description: Any AEs including SAEs that lead to withdrawal from the study are considered under this outcome measure.
  A participant is considered to have withdrawn from the study if no new study procedure has been performed or no new information has been collected for him/her since the date of withdrawal/last contact.
Time Frame: From Day 1 to Day 197
Population: The analysis was performed on the exposed set. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 12 | 24 | 24 | 24
Participants | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With SAEs Leading to Withholding Further Study Intervention Administration
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, results in abnormal pregnancy outcomes or any other situation based on appropriate medical or scientific judgement.
  SAEs that lead to withholding of the study intervention administration were considered under this outcome measure.
Time Frame: From Day 1 to Day 197
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 12 | 24 | 24 | 24
Participants | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With AEs Leading to Withholding Further Study Intervention Administration
Description: An AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention.
  AEs that lead to withholding of the study intervention administration were considered under this outcome measure.
Time Frame: From Day 1 to Day 197
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 12 | 24 | 24 | 24
Participants | 0 | 1 | 1 | 0 | 1

11. Primary Outcome: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 8
Description: Assessed hematological laboratory parameters include basophils, eosinophils, erythrocytes, hemoglobin, hematocrit, lymphocytes, monocytes, neutrophils, platelets, leukocytes. Hepatic laboratory parameters include alanine aminotransferase [ALT], aspartate aminotransferase [AST] and renal laboratory parameters include creatinine and blood urea. Categories reported when comparing Day 1 (baseline) and Day 8 hematological, renal and hepatic laboratory results are defined as follows: <parameter>-<range at baseline>-<range at timing> (e.g. ALT-Within-Within). Range level being classified as below, within or above the normal range.
Time Frame: At Day 8 compared to Day 1 (Baseline)
Population: The analysis was performed on the exposed set. Only participants with data available at the mentioned timepoints were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 12 | 24 | 24 | 24
Participants
  ALT-Below -Below | 0 | 0 | 0 | 0 | 0
  ALT-Within-Below | 0 | 0 | 0 | 0 | 0
  ALT-Above-Below | 0 | 0 | 0 | 0 | 0
  ALT-Below-Within | 0 | 0 | 0 | 0 | 0
  ALT-Within-Within | 11 | 11 | 23 | 23 | 24
  ALT-Above-Within | 0 | 0 | 0 | 1 | 0
  ALT-Below-Above | 0 | 0 | 0 | 0 | 0
  ALT-Within-Above | 1 | 0 | 0 | 0 | 0
  ALT-Above-Above | 0 | 1 | 0 | 0 | 0
  AST-Below-Below | 0 | 0 | 0 | 0 | 0
  AST-Within-Below | 0 | 0 | 0 | 0 | 0
  AST-Above-Below | 0 | 0 | 0 | 0 | 0
  AST-Below-Within | 0 | 0 | 0 | 0 | 0
  AST-Within-Within | 12 | 12 | 23 | 22 | 23
  AST-Above-Within | 0 | 0 | 0 | 2 | 1
  AST-Below-Above | 0 | 0 | 0 | 0 | 0
  AST-Within-Above | 0 | 0 | 0 | 0 | 0
  AST-Above-Above | 0 | 0 | 0 | 0 | 0
  Creatinine-Below-Below | 0 | 0 | 0 | 0 | 0
  Creatinine-Within-Below | 0 | 1 | 0 | 0 | 0
  Creatinine-Above-Below | 0 | 0 | 0 | 0 | 0
  Creatinine-Below-Within | 0 | 0 | 0 | 0 | 0
  Creatinine-Within-Within | 11 | 10 | 21 | 22 | 20
  Creatinine-Above-Within | 0 | 0 | 2 | 2 | 1
  Creatinine-Below-Above | 0 | 0 | 0 | 0 | 0
  Creatinine-Within-Above | 1 | 0 | 0 | 0 | 0
  Creatinine-Above-Above | 0 | 1 | 0 | 0 | 3
  Blood urea-Below-Below | 0 | 0 | 1 | 1 | 0
  Blood urea-Within-Below | 0 | 1 | 2 | 0 | 0
  Blood urea-Above-Below | 0 | 0 | 0 | 0 | 0
  Blood urea-Below-Within | 1 | 1 | 0 | 3 | 0
  Blood urea-Within-Within | 11 | 10 | 20 | 20 | 24
  Blood urea-Above-Within | 0 | 0 | 0 | 0 | 0
  Blood urea-Below-Above | 0 | 0 | 0 | 0 | 0
  Blood urea-Within-Above | 0 | 0 | 0 | 0 | 0
  Blood urea-Above-Above | 0 | 0 | 0 | 0 | 0
  Basophils-Below-Below | 0 | 0 | 0 | 0 | 0
  Basophils-Within-Below | 0 | 0 | 0 | 0 | 0
  Basophils-Above-Below | 0 | 0 | 0 | 0 | 0
  Basophils-Below-Within | 0 | 0 | 0 | 0 | 0
  Basophils-Within-Within | 12 | 10 | 23 | 24 | 24
  Basophils-Above-Within | 0 | 0 | 0 | 0 | 0
  Basophils-Below-Above | 0 | 0 | 0 | 0 | 0
  Basophils-Within-Above | 0 | 1 | 0 | 0 | 0
  Basophils-Above-Above | 0 | 0 | 0 | 0 | 0
  Eosinophils-Below-Below | 0 | 0 | 0 | 0 | 0
  Eosinophils-Within-Below | 0 | 0 | 0 | 0 | 0
  Eosinophils-Above-Below | 0 | 0 | 0 | 0 | 0
  Eosinophils-Below-Within | 0 | 0 | 0 | 0 | 0
  Eosinophils-Within-Within | 12 | 10 | 21 | 24 | 24
  Eosinophils-Above-Within | 0 | 0 | 0 | 0 | 0
  Eosinophils-Below-Above | 0 | 0 | 0 | 0 | 0
  Eosinophils-Within-Above | 0 | 0 | 0 | 0 | 0
  Eosinophils-Above-Above | 0 | 1 | 2 | 0 | 0
  Hematocrit-Below-Below | 0 | 0 | 0 | 0 | 0
  Hematocrit-Within-Below | 0 | 0 | 0 | 0 | 0
  Hematocrit-Above-Below | 0 | 0 | 0 | 0 | 0
  Hematocrit-Below-Within | 0 | 0 | 0 | 0 | 1
  Hematocrit-Within-Within | 12 | 12 | 22 | 22 | 23
  Hematocrit-Above-Within | 0 | 0 | 1 | 1 | 0
  Hematocrit-Below-Above | 0 | 0 | 0 | 0 | 0
  Hematocrit-Within-Above | 0 | 0 | 0 | 1 | 0
  Hematocrit-Above-Above | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Below-Below | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Within-Below | 0 | 0 | 2 | 0 | 0
  Hemoglobin-Above-Below | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Below-Within | 0 | 0 | 0 | 0 | 2
  Hemoglobin-Within-Within | 12 | 12 | 21 | 23 | 22
  Hemoglobin-Above-Within | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Below-Above | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Within-Above | 0 | 0 | 0 | 1 | 0
  Hemoglobin-Above-Above | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Below-Below | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Within-Below | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Above-Below | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Below-Within | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Within-Within | 10 | 11 | 22 | 24 | 24
  Lymphocytes-Above-Within | 1 | 0 | 0 | 0 | 0
  Lymphocytes-Below-Above | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Within-Above | 1 | 0 | 1 | 0 | 0
  Lymphocytes-Above-Above | 0 | 0 | 0 | 0 | 0
  Monocytes-Below-Below | 0 | 0 | 0 | 0 | 0
  Monocytes-Within-Below | 1 | 0 | 0 | 0 | 0
  Monocytes-Above-Below | 0 | 0 | 0 | 0 | 0
  Monocytes-Below-Within | 0 | 0 | 0 | 1 | 0
  Monocytes-Within-Within | 11 | 11 | 23 | 23 | 23
  Monocytes-Above-Within | 0 | 0 | 0 | 0 | 1
  Monocytes-Below-Above | 0 | 0 | 0 | 0 | 0
  Monocytes-Within-Above | 0 | 0 | 0 | 0 | 0
  Monocytes-Above-Above | 0 | 0 | 0 | 0 | 0
  Neutrophils-Below-Below | 0 | 0 | 0 | 0 | 0
  Neutrophils-Within-Below | 0 | 0 | 0 | 0 | 0
  Neutrophils-Above-Below | 0 | 0 | 0 | 0 | 0
  Neutrophils-Below-Within | 0 | 1 | 0 | 0 | 0
  Neutrophils-Within-Within | 12 | 10 | 20 | 22 | 24
  Neutrophils-Above-Within | 0 | 0 | 1 | 1 | 0
  Neutrophils-Below-Above | 0 | 0 | 0 | 0 | 0
  Neutrophils-Within-Above | 0 | 0 | 2 | 1 | 0
  Neutrophils-Above-Above | 0 | 0 | 0 | 0 | 0
  Platelets-Below-Below | 0 | 0 | 0 | 0 | 0
  Platelets-Within-Below | 0 | 0 | 0 | 0 | 0
  Platelets-Above-Below | 0 | 0 | 0 | 0 | 0
  Platelets-Below-Within | 0 | 0 | 0 | 0 | 0
  Platelets-Within-Within | 10 | 11 | 21 | 22 | 23
  Platelets-Above-Within | 1 | 0 | 0 | 1 | 1
  Platelets-Below-Above | 0 | 0 | 0 | 0 | 0
  Platelets-Within-Above | 0 | 1 | 1 | 0 | 0
  Platelets-Above-Above | 1 | 0 | 1 | 1 | 0
  Erythrocytes-Below-Below | 0 | 0 | 0 | 0 | 0
  Erythrocytes-Within-Below | 0 | 0 | 0 | 1 | 0
  Erythrocytes-Above-Below | 0 | 0 | 0 | 0 | 0
  Erythrocytes-Below-Within | 0 | 0 | 0 | 0 | 0
  Erythrocytes-Within-Within | 12 | 12 | 23 | 21 | 24
  Erythrocytes-Above-Within | 0 | 0 | 0 | 1 | 0
  Erythrocytes-Below-Above | 0 | 0 | 0 | 0 | 0
  Erythrocytes-Within-Above | 0 | 0 | 0 | 1 | 0
  Erythrocytes-Above-Above | 0 | 0 | 0 | 0 | 0
  Leukocytes-Below-Below | 0 | 1 | 0 | 0 | 0
  Leukocytes-Within-Below | 2 | 0 | 0 | 0 | 0
  Leukocytes-Above-Below | 0 | 0 | 0 | 0 | 0
  Leukocytes-Below-Within | 0 | 1 | 0 | 1 | 2
  Leukocytes-Within-Within | 9 | 10 | 21 | 23 | 22
  Leukocytes-Above-Within | 0 | 0 | 1 | 0 | 0
  Leukocytes-Below-Above | 0 | 0 | 0 | 0 | 0
  Leukocytes-Within-Above | 1 | 0 | 1 | 0 | 0
  Leukocytes-Above-Above | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Deviations From Normal or Baseline Values of Haematological, Renal, and Hepatic Panel Test Results at Day 176
Description: Assessed hematological laboratory parameters include basophils, eosinophils, erythrocytes, hemoglobin, hematocrit, lymphocytes, monocytes, neutrophils, platelets, leukocytes. Hepatic laboratory parameters include alanine aminotransferase [ALT], aspartate aminotransferase [AST] and renal laboratory parameters include creatinine and blood urea. Categories reported when comparing Day 169 (baseline) and Day 176 hematological, renal and hepatic laboratory results are defined as follows: <parameter>-<range at baseline>-<range at timing> (e.g. ALT-Within-Within). Range level being classified as below, within or above the normal range.
Time Frame: At Day 176 compared to Day 169 (Baseline)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 8 | 10 | 21 | 22 | 21
Participants
  ALT-Below-Below | 0 | 0 | 0 | 0 | 0
  ALT-Within-Below | 0 | 0 | 0 | 0 | 0
  ALT-Above-Below | 0 | 0 | 0 | 0 | 0
  ALT-Below-Within | 0 | 0 | 0 | 0 | 0
  ALT-Within-Within | 7 | 10 | 20 | 20 | 20
  ALT-Above-Within | 1 | 0 | 0 | 1 | 1
  ALT-Below-Above | 0 | 0 | 0 | 0 | 0
  ALT-Within-Above | 0 | 0 | 1 | 0 | 0
  ALT-Above-Above | 0 | 0 | 0 | 1 | 0
  AST-Below-Below | 0 | 0 | 0 | 0 | 0
  AST-Within-Below | 0 | 0 | 0 | 0 | 0
  AST-Above-Below | 0 | 0 | 0 | 0 | 0
  AST-Below-Within | 0 | 0 | 0 | 0 | 0
  AST-Within-Within | 7 | 10 | 19 | 20 | 20
  AST-Above-Within | 1 | 0 | 0 | 0 | 0
  AST-Below-Above | 0 | 0 | 0 | 0 | 0
  AST-Within-Above | 0 | 0 | 2 | 2 | 1
  AST-Above-Above | 0 | 0 | 0 | 0 | 0
  Creatinine-Below-Below | 0 | 2 | 0 | 0 | 0
  Creatinine-Within-Below | 0 | 0 | 0 | 0 | 0
  Creatinine-Above-Below | 0 | 0 | 0 | 0 | 0
  Creatinine-Below-Within | 0 | 0 | 0 | 0 | 0
  Creatinine-Within-Within | 8 | 7 | 18 | 19 | 18
  Creatinine-Above-Within | 0 | 0 | 2 | 1 | 1
  Creatinine-Below-Above | 0 | 0 | 0 | 0 | 0
  Creatinine-Within-Above | 0 | 0 | 1 | 1 | 1
  Creatinine-Above-Above | 0 | 1 | 0 | 1 | 1
  Blood urea-Below-Below | 0 | 0 | 0 | 0 | 0
  Blood urea-Within-Below | 1 | 0 | 0 | 0 | 1
  Blood urea-Above-Below | 0 | 0 | 0 | 0 | 0
  Blood urea-Below-Within | 1 | 0 | 1 | 0 | 1
  Blood urea-Within-Within | 6 | 10 | 20 | 22 | 19
  Blood urea-Above-Within | 0 | 0 | 0 | 0 | 0
  Blood urea-Below-Above | 0 | 0 | 0 | 0 | 0
  Blood urea-Within-Above | 0 | 0 | 0 | 0 | 0
  Blood urea-Above-Above | 0 | 0 | 0 | 0 | 0
  Basophils-Below-Below | 0 | 0 | 0 | 0 | 0
  Basophils-Within-Below | 0 | 0 | 0 | 0 | 0
  Basophils-Above-Below | 0 | 0 | 0 | 0 | 0
  Basophils-Below-Within | 0 | 0 | 0 | 0 | 0
  Basophils-Within-Within | 8 | 10 | 21 | 22 | 21
  Basophils-Above-Within | 0 | 0 | 0 | 0 | 0
  Basophils-Below-Above | 0 | 0 | 0 | 0 | 0
  Basophils-Within-Above | 0 | 0 | 0 | 0 | 0
  Basophils-Above-Above | 0 | 0 | 0 | 0 | 0
  Eosinophils-Below-Below | 0 | 0 | 0 | 0 | 0
  Eosinophils-Within-Below | 0 | 0 | 0 | 0 | 0
  Eosinophils-Above-Below | 0 | 0 | 0 | 0 | 0
  Eosinophils-Below-Within | 0 | 0 | 0 | 0 | 0
  Eosinophils-Within-Within | 7 | 10 | 20 | 22 | 21
  Eosinophils-Above-Within | 0 | 0 | 1 | 0 | 0
  Eosinophils-Below-Above | 0 | 0 | 0 | 0 | 0
  Eosinophils-Within-Above | 1 | 0 | 0 | 0 | 0
  Eosinophils-Above-Above | 0 | 0 | 0 | 0 | 0
  Hematocrit-Below-Below | 0 | 0 | 0 | 0 | 0
  Hematocrit-Within-Below | 0 | 0 | 0 | 0 | 0
  Hematocrit-Above-Below | 0 | 0 | 0 | 0 | 0
  Hematocrit-Below-Within | 0 | 0 | 0 | 0 | 0
  Hematocrit-Within-Within | 8 | 10 | 18 | 22 | 20
  Hematocrit-Above-Within | 0 | 0 | 1 | 0 | 1
  Hematocrit-Below-Above | 0 | 0 | 0 | 0 | 0
  Hematocrit-Within-Above | 0 | 0 | 2 | 0 | 0
  Hematocrit-Above-Above | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Below-Below | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Within-Below | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Above-Below | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Below-Within | 0 | 0 | 0 | 1 | 1
  Hemoglobin-Within-Within | 8 | 10 | 21 | 21 | 20
  Hemoglobin-Above-Within | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Below-Above | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Within-Above | 0 | 0 | 0 | 0 | 0
  Hemoglobin-Above-Above | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Below-Below | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Within-Below | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Above-Below | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Below-Within | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Within-Within | 8 | 10 | 20 | 22 | 21
  Lymphocytes-Above-Within | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Below-Above | 0 | 0 | 0 | 0 | 0
  Lymphocytes-Within-Above | 0 | 0 | 1 | 0 | 0
  Lymphocytes-Above-Above | 0 | 0 | 0 | 0 | 0
  Monocytes-Below-Below | 0 | 0 | 0 | 0 | 0
  Monocytes-Within-Below | 0 | 0 | 0 | 0 | 0
  Monocytes-Above-Below | 0 | 0 | 0 | 0 | 0
  Monocytes-Below-Within | 0 | 0 | 0 | 0 | 0
  Monocytes-Within-Within | 8 | 10 | 21 | 22 | 21
  Monocytes-Above-Within | 0 | 0 | 0 | 0 | 0
  Monocytes-Below-Above | 0 | 0 | 0 | 0 | 0
  Monocytes-Within-Above | 0 | 0 | 0 | 0 | 0
  Monocytes-Above-Above | 0 | 0 | 0 | 0 | 0
  Neutrophils-Below-Below | 0 | 0 | 0 | 0 | 0
  Neutrophils-Within-Below | 0 | 0 | 0 | 0 | 0
  Neutrophils-Above-Below | 0 | 0 | 0 | 0 | 0
  Neutrophils-Below-Within | 0 | 0 | 0 | 0 | 0
  Neutrophils-Within-Within | 8 | 10 | 18 | 22 | 15
  Neutrophils-Above-Within | 0 | 0 | 2 | 0 | 6
  Neutrophils-Below-Above | 0 | 0 | 0 | 0 | 0
  Neutrophils-Within-Above | 0 | 0 | 1 | 0 | 0
  Neutrophils-Above-Above | 0 | 0 | 0 | 0 | 0
  Platelets-Below-Below | 0 | 0 | 0 | 0 | 0
  Platelets-Within-Below | 0 | 0 | 0 | 1 | 0
  Platelets-Above-Below | 0 | 0 | 0 | 0 | 0
  Platelets-Below-Within | 0 | 0 | 0 | 0 | 0
  Platelets-Within-Within | 8 | 10 | 19 | 21 | 20
  Platelets-Above-Within | 0 | 0 | 2 | 0 | 1
  Platelets-Below-Above | 0 | 0 | 0 | 0 | 0
  Platelets-Within-Above | 0 | 0 | 0 | 0 | 0
  Platelets-Above-Above | 0 | 0 | 0 | 0 | 0
  Erythrocytes-Below-Below | 0 | 0 | 0 | 0 | 0
  Erythrocytes-Within-Below | 0 | 0 | 0 | 0 | 0
  Erythrocytes-Above-Below | 0 | 0 | 0 | 0 | 0
  Erythrocytes-Below-Within | 0 | 0 | 0 | 1 | 1
  Erythrocytes-Within-Within | 8 | 10 | 21 | 20 | 19
  Erythrocytes-Above-Within | 0 | 0 | 0 | 1 | 1
  Erythrocytes-Below-Above | 0 | 0 | 0 | 0 | 0
  Erythrocytes-Within-Above | 0 | 0 | 0 | 0 | 0
  Erythrocytes-Above-Above | 0 | 0 | 0 | 0 | 0
  Leukocytes-Below-Below | 0 | 0 | 0 | 0 | 0
  Leukocytes-Within-Below | 0 | 0 | 0 | 0 | 0
  Leukocytes-Above-Below | 0 | 0 | 0 | 0 | 0
  Leukocytes-Below-Within | 0 | 0 | 1 | 0 | 1
  Leukocytes-Within-Within | 8 | 10 | 18 | 22 | 19
  Leukocytes-Above-Within | 0 | 0 | 2 | 0 | 1
  Leukocytes-Below-Above | 0 | 0 | 0 | 0 | 0
  Leukocytes-Within-Above | 0 | 0 | 0 | 0 | 0
  Leukocytes-Above-Above | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Any SAE
Description: as for outcome 7
Time Frame: From Day 197 to Day 337
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 12 | 24 | 24 | 24
Participants | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With AEs/SAEs Leading to Withdrawal From the Study
Description: as for outcome 8
Time Frame: From Day 197 to Day 337
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 12 | 24 | 24 | 24
Participants | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Anti-Vi Antigen Immunoglobulin G (IgG) Antibody Concentrations
Description: Anti-Vi specific IgG antibodies were measured by an anti-Vi IgG Enzyme-Linked Immunosorbent Assay (ELISA) kit. Blood samples were collected at specified timepoints.
Time Frame: At Day 1 (pre-dose 1), Day 29, Day 169 (pre-Dose 2), Day 176 and Day 197
Population: The analysis was performed on Per-protocol set, which included all eligible participants who received each dose as per-protocol, had immunogenicity results post- dose, complied with dosing/blood draw intervals, without intercurrent conditions that may interfere with immunogenicity and without prohibited concomitant medication/vaccination during the specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (µg/mL)
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 11 | 21 | 24 | 24
microgram per milliliter (µg/mL)
  Day 1 (pre-dose 1) | 1.10 [NA to NA] — 95% CI are not applicable for GMCs at Day 1 when all participants were below LLOQ (lower limit of quantification) | 1.52 [0.93 to 2.48] | 1.14 [1.06 to 1.23] | 1.17 [1.03 to 1.33] | 1.10 [NA to NA] — 95% CI are not applicable for GMCs at Day 1 when all participants were below LLOQ
  Day 29 | 14.12 [8.21 to 24.29] | 19.61 [9.10 to 42.28] | 60.52 [35.28 to 103.82] | 36.97 [20.56 to 66.48] | 4.95 [3.23 to 7.59]
  Day 169 (pre-Dose 2): number analyzed (Participants) | 8 | 10 | 21 | 22 | 21
  Day 169 (pre-Dose 2) | 4.36 [2.01 to 9.47] | 11.17 [4.79 to 26.03] | 18.58 [9.97 to 34.60] | 12.55 [7.06 to 22.32] | 6.18 [3.50 to 10.92]
  Day 176: number analyzed (Participants) | 8 | 10 | 18 | 18 | 19
  Day 176 | 10.90 [4.72 to 25.21] | 18.78 [9.05 to 38.97] | 32.38 [19.82 to 52.89] | 56.78 [38.23 to 84.32] | 5.15 [3.02 to 8.77]
  Day 197: number analyzed (Participants) | 8 | 8 | 16 | 18 | 20
  Day 197 | 10.16 [5.08 to 20.30] | 18.88 [8.23 to 43.29] | 33.75 [17.78 to 64.07] | 37.14 [23.79 to 58.00] | 5.17 [3.14 to 8.52]

16. Secondary Outcome: Geometric Mean Ratio (GMR) for Anti-Vi Antigen IgG Antibody Concentrations
Description: Anti-Vi specific IgG antibodies were measured by an anti-Vi IgG ELISA kit. Blood samples were collected at specified timepoints. Within participant GMRs were calculated as ratio of concentration in the post-vaccination timepoint to the pre-vaccination timepoint.
Time Frame: At Day 29, Day 169, Day 176, and Day 197 compared to Day 1 (baseline)
Population: The analysis was performed on the Per-protocol set. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 11 | 21 | 24 | 24
Ratio
  Day 29 | 12.84 [7.46 to 22.08] | 12.90 [6.77 to 24.58] | 53.01 [31.94 to 87.99] | 31.55 [18.74 to 53.11] | 4.50 [2.93 to 6.90]
  Day 169: number analyzed (Participants) | 8 | 10 | 21 | 22 | 21
  Day 169 | 3.96 [1.82 to 8.61] | 7.11 [3.51 to 14.40] | 16.27 [8.94 to 29.61] | 10.65 [6.59 to 17.22] | 5.62 [3.18 to 9.93]
  Day 176: number analyzed (Participants) | 8 | 10 | 18 | 18 | 19
  Day 176 | 9.91 [4.29 to 22.92] | 11.96 [6.05 to 23.65] | 28.19 [17.72 to 44.84] | 47.45 [36.38 to 61.89] | 4.68 [2.75 to 7.97]
  Day 197: number analyzed (Participants) | 8 | 8 | 16 | 18 | 20
  Day 197 | 9.23 [4.62 to 18.46] | 11.00 [5.15 to 23.49] | 29.22 [15.71 to 54.35] | 31.04 [23.14 to 41.65] | 4.70 [2.85 to 7.74]

17. Secondary Outcome: GMR for Anti-Vi Antigen IgG Antibody Concentrations
Description: as for outcome 16
Time Frame: At Day 176 and Day 197 compared to Day 169 (baseline)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 8 | 10 | 18 | 18 | 20
Ratio
  Day 176: number analyzed (Participants) | 8 | 10 | 18 | 18 | 19
  Day 176 | 2.50 [1.63 to 3.83] | 1.68 [1.16 to 2.43] | 2.00 [1.06 to 3.80] | 4.20 [2.46 to 7.17] | 0.82 [0.47 to 1.43]
  Day 197: number analyzed (Participants) | 8 | 8 | 16 | 18 | 20
  Day 197 | 2.33 [1.67 to 3.25] | 1.72 [1.17 to 2.54] | 1.71 [1.21 to 2.43] | 3.08 [2.09 to 4.53] | 0.77 [0.45 to 1.31]

18. Secondary Outcome: GMC of Anti-O:2 IgG Antibody Concentrations
Description: Anti-O:2 IgG antibodies in serum were measured by an ELISA assay. Blood samples were collected at specified timepoints.
Time Frame: At Day 1 (pre-dose 1), Day 29, Day 169 (pre-dose 2), Day 176 and Day 197
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Units per milliliter (EU/mL)
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 11 | 21 | 24 | 24
ELISA Units per milliliter (EU/mL)
  Day 1 (pre-dose 1) | 36.35 [15.21 to 86.89] | 28.31 [11.29 to 70.97] | 25.28 [14.73 to 43.39] | 25.90 [13.56 to 49.44] | 22.15 [13.18 to 37.23]
  Day 29 | 4150.79 [1362.97 to 12640.82] | 559.62 [177.08 to 1768.50] | 4110.58 [1975.76 to 8552.10] | 668.30 [314.08 to 1422.01] | 28.19 [16.07 to 49.47]
  Day 169 (pre-dose 2): number analyzed (Participants) | 8 | 10 | 21 | 22 | 21
  Day 169 (pre-dose 2) | 702.49 [138.39 to 3565.88] | 298.02 [85.01 to 1044.76] | 894.08 [397.22 to 2012.40] | 268.09 [124.74 to 576.18] | 18.43 [10.91 to 31.13]
  Day 176: number analyzed (Participants) | 8 | 10 | 18 | 18 | 19
  Day 176 | 1079.75 [322.08 to 3619.77] | 464.70 [188.39 to 1146.25] | 1342.38 [644.96 to 2793.95] | 522.60 [264.74 to 1031.60] | 18.24 [10.38 to 32.05]
  Day 197: number analyzed (Participants) | 8 | 8 | 16 | 18 | 20
  Day 197 | 958.21 [298.69 to 3074.02] | 520.77 [167.69 to 1617.23] | 956.89 [440.21 to 2080.03] | 388.50 [219.98 to 686.13] | 17.28 [10.13 to 29.47]

19. Secondary Outcome: GMR for Anti-O:2 IgG Antibody Concentrations
Description: Anti-O:2 IgG antibodies in serum were measured by an ELISA assay. Blood samples were collected at specified timepoints. Within participant GMRs were calculated as ratio of concentration in the post-vaccination timepoint to the pre-vaccination timepoint.
Time Frame: At Day 29, Day 169, Day 176, and Day 197 compared to Day 1 (baseline)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 11 | 21 | 24 | 24
Ratio
  Day 29 | 114.19 [44.83 to 290.86] | 19.77 [10.03 to 38.96] | 162.61 [91.17 to 290.04] | 25.81 [13.15 to 50.64] | 1.27 [1.02 to 1.60]
  Day 169: number analyzed (Participants) | 8 | 10 | 21 | 22 | 21
  Day 169 | 26.15 [6.12 to 111.64] | 9.11 [3.83 to 21.64] | 37.28 [20.47 to 67.89] | 9.15 [4.52 to 18.51] | 0.92 [0.80 to 1.07]
  Day 176: number analyzed (Participants) | 8 | 10 | 18 | 18 | 19
  Day 176 | 40.19 [11.79 to 136.94] | 14.20 [7.11 to 28.38] | 68.01 [39.46 to 117.23] | 19.12 [8.97 to 40.76] | 0.86 [0.77 to 0.96]
  Day 197: number analyzed (Participants) | 8 | 8 | 16 | 18 | 20
  Day 197 | 35.66 [10.36 to 122.82] | 19.23 [9.58 to 38.60] | 51.16 [27.32 to 95.79] | 17.86 [9.42 to 33.86] | 0.95 [0.81 to 1.12]

20. Secondary Outcome: GMR for Anti-O:2 IgG Antibody Concentrations
Description: Anti-O:2 IgG antibodies in serum were measured by an ELISA assay. Blood samples were collected at specified timepoint. Within participant GMRs were calculated as ratio of concentration in the post-vaccination timepoint to the pre-vaccination timepoint.
Time Frame: At Day 176 and Day 197 compared to Day 169 (baseline)
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 8 | 10 | 18 | 18 | 20
Ratio
  Day 176: number analyzed (Participants) | 8 | 10 | 18 | 18 | 19
  Day 176 | 1.54 [0.82 to 2.88] | 1.56 [1.07 to 2.28] | 1.76 [1.31 to 2.36] | 1.89 [1.34 to 2.67] | 0.98 [0.92 to 1.04]
  Day 197: number analyzed (Participants) | 8 | 8 | 16 | 18 | 20
  Day 197 | 1.36 [0.67 to 2.76] | 1.70 [0.90 to 3.22] | 1.60 [1.23 to 2.09] | 2.01 [1.42 to 2.84] | 0.99 [0.92 to 1.07]

21. Secondary Outcome: Number of Participants With Anti-Vi Antigen IgG Antibody Concentrations Greater Than or Equal to (>=) 4.3 Micrograms Per Milliliter (µg/mL)
Description: Blood samples were collected at specified timepoint for each component as measured by ELISA.
Time Frame: At Day 1, Day 29, Day 169, Day 176 and Day 197
Population: The analysis was performed on Full Analysis Set (FAS), which included all participants who received at least 1 dose of the study intervention and had post- vaccination immunogenicity data during the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 11 | 22 | 24 | 24
Participants
  Day 1 | 0 | 2 | 0 | 1 | 0
  Day 29 | 12 | 10 | 22 | 23 | 13
  Day 169: number analyzed (Participants) | 8 | 11 | 21 | 22 | 21
  Day 169 | 6 | 10 | 20 | 18 | 13
  Day 176: number analyzed (Participants) | 8 | 10 | 20 | 21 | 21
  Day 176 | 6 | 9 | 19 | 21 | 12
  Day 197: number analyzed (Participants) | 8 | 10 | 21 | 22 | 21
  Day 197 | 7 | 9 | 20 | 22 | 12

22. Secondary Outcome: Number of Participants With Anti-Vi Antigen IgG Antibody Concentrations >= 2.0 µg/mL
Description: Blood samples were collected at specified timepoint for each component as measured by ELISA.
Time Frame: At Day 1, Day 29, Day 169, Day 176 and Day 197
Population: The analysis was performed on FAS. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 11 | 22 | 24 | 24
Participants
  Day 1 | 0 | 2 | 1 | 1 | 0
  Day 29 | 12 | 11 | 22 | 23 | 20
  Day 169: number analyzed (Participants) | 8 | 11 | 21 | 22 | 21
  Day 169 | 6 | 10 | 20 | 22 | 17
  Day 176: number analyzed (Participants) | 8 | 10 | 20 | 21 | 21
  Day 176 | 8 | 10 | 19 | 21 | 16
  Day 197: number analyzed (Participants) | 8 | 10 | 21 | 22 | 21
  Day 197 | 8 | 10 | 21 | 22 | 16

23. Secondary Outcome: Number of Participants With at Least 4-fold Increase in Anti-O:2 IgG Antibody Concentrations
Description: Blood samples were collected at specified timepoint for each component as measured by ELISA. 4-fold increase was defined as 4 times the baseline value of anti-O:2 IgG antibody concentrations.
Time Frame: At Day 29, Day 169, Day 176 and Day 197 compared to Day 1 (baseline)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
Number analyzed (Participants) | 12 | 11 | 22 | 24 | 24
Participants
  Day 29 | 12 | 9 | 22 | 20 | 1
  Day 169: number analyzed (Participants) | 8 | 11 | 21 | 22 | 21
  Day 169 | 7 | 7 | 20 | 16 | 0
  Day 176: number analyzed (Participants) | 8 | 10 | 20 | 21 | 21
  Day 176 | 8 | 8 | 20 | 18 | 0
  Day 197: number analyzed (Participants) | 8 | 10 | 21 | 22 | 21
  Day 197 | 8 | 9 | 20 | 19 | 0

ADVERSE EVENTS:
Time Frame: SAEs were reported from Day 1 to Day 337 (end of study), solicited AEs were reported from Day 1 to Day 7 and Day 169 to Day 175, and unsolicited AEs were reported from Day 1 to Day 28 and Day 169 to Day 196. Laboratory abnormalities were reported as change from baseline (Day 1[first dose] and Day 169 [second dose]) to 7 days post-vaccination (Day 8, and Day 176 respectively).
Description: SAEs, solicited AEs and unsolicited AEs were reported for the Exposed set. Exposed set included all participants who received at least 1 dose of the study intervention.
Arm/Group | Step 1a: Low Dose TYP04A Vaccine Without Alum | Step 1b: Low Dose TYP03A Vaccine With Alum | Step 2: Full Dose TYP04B Vaccine Without Alum | Step 2: Full Dose TYP03B Vaccine With Alum | Control: TYPHIM VI and BOOSTRIX Vaccine
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 9/12 | 12/12 | 24/24 | 24/24 | 24/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Step 1a: Low Dose TYP04A Vaccine Without Alum (N=12) | Step 1b: Low Dose TYP03A Vaccine With Alum (N=12) | Step 2: Full Dose TYP04B Vaccine Without Alum (N=24) | Step 2: Full Dose TYP03B Vaccine With Alum (N=24) | Control: TYPHIM VI and BOOSTRIX Vaccine (N=24)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thyroid calcification (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Administration site erythema (General disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Administration site pain (General disorders) | 6 (9) | 11 (17) | 21 (40) | 23 (41) | 22 (30)
Administration site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Administration site swelling (General disorders) | 1 (2) | 0 (0) | 3 (3) | 1 (2) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (5) | 5 (6) | 11 (15) | 15 (22) | 15 (21)
Hangover (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site movement impairment (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site movement impairment (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (4) | 3 (3) | 5 (5) | 5 (5)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 3 (4) | 0 (0) | 0 (0)
Extraskeletal ossification (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Human papilloma virus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 4 (4) | 3 (5) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (6) | 12 (16) | 16 (24) | 13 (18)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (7) | 6 (9) | 14 (21) | 11 (15) | 17 (26)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcoholic hangover (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethritis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT05613205/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT05613205/SAP_001.pdf